CLINICAL TRIAL: NCT00167856
Title: Effects of Venlafaxine on Chronic Neuropathic Pain Following Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Widerstrom-Noga, Eva - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: B3070-R
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2009-02

CONDITIONS: Neuropathic Pain; Pain; Spinal Cord Injuries
Keywords: Burning pain; Clinical trial; Effexor; Pain; Spinal cord injury; Venalafaxine; Neuropathic Pain
MeSH Terms: conditions — Neuralgia; Pain; Spinal Cord Injuries | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Venlafaxine HCL (extended release)
  Interventions: Drug: Venalafaxine hydrochloride
- 2 (Active Comparator): Benztropine Mesylate
  Interventions: Drug: Venalafaxine hydrochloride

INTERVENTIONS:
Drug: Venalafaxine hydrochloride — Norepinephrine/Serotonin Reuptake Inhibitor (NSRI)
  Other Names: Effexor XR

SUMMARY:
The purpose of this study is to evaluate the pain-relieving effects of venlafaxine hydrochloride (Effexor) in chronic neuropathic (burning, shock-like, electric) pain after spinal cord injury (SCI). Although a number of medications have been used to treat SCI pain, no drug has been consistently helpful, and, therefore, many people with SCI continue to have difficult chronic pain. Venlafaxine is a new anti-depressant drug that has not been tested for use in SCI neuropathic pain, but has been helpful for other types of neuropathic pain.

DETAILED DESCRIPTION:
Persistent pain is one of the most common reasons for impaired quality of life following spinal cord injury (SCI). Although numerous interventions are often used to manage neuropathic pain following SCI, most people receive inadequate relief and continue to suffer many years after the original injury. The long-term goal of our pain research is to improve the management of chronic neuropathic pain following SCI.

This study examines the effect of Venlafaxine hydrochloride (VH) in the treatment of chronic neuropathic pain associated with SCI. VH is a second-generation, structurally novel antidepressant medication with a mild side-effect profile compared to these older tricyclic antidepressants (e.g. imipramine and amitriptyline). Previous clinical trials suggest that approximately 60-70% of people with heterogeneous neuropathic pain report at least moderate reductions in pain with older antidepressants. However, reported side-effects have been numerous, and few trials have been conducted on neuropathic pain due to SCI.

The current study is a two-period, 24-week crossover, randomized, placebo-controlled trial. A sample of 60 persons with chronic neuropathic pain and SCI will be randomly assigned to either of two treatment groups (n=30 for each group), in a double-blind fashion. One group will receive VH first and then placebo, whereas the second group will start with the placebo followed by the VH. There will be weekly contacts between the research staff and the study participants to assess pain relief and medication side effects (presence and severity). Several measures of pain intensity, psychosocial well-being, quality of life, and sensory function will be taken throughout the study to examine the effects of VH on neuropathic pain.

We expect that VH will help to relieve neuropathic pain in persons with SCI, and that this decrease in pain intensity will correlate with a reduced psychosocial impact, improved mood, increased participation in daily activities, and increased life satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* participant must be able to swallow pills
* fluent in English
* incomplete or complete spinal cord injury
* presence of at least moderately severe neuropathic pain at or below the level of injury
* spinal cord injury at least 2 year prior to entering the study
* pain for at least 6 months prior to entering the study
* spinal cord injury level above L1
* participants on anticonvulsants are considered
* approval of primary physician

Exclusion Criteria:

* pregnant women, or those contemplating pregnancy
* prior history of use of Venlafaxine hydrochloride (Effexor)
* current use of MAOI medications
* persons who have a recent (past year) history of alcohol or drug abuse
* persons with a history of renal disease, heart disease or uncontrolled hypertension, liver disease or hepatic cirrhosis, active major medical or psychiatric illness
* persons with a significant post-traumatic encephalopathy from head trauma sustained at SCI
* persons with tardive dyskinesia or narrow angle glaucoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-06; Primary Completion 2007-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Pain Intensity as measured by subject pain diaries | Baseline (2 Weeks); Phase 1 (1 week at max dose); Washout (2 weeks); Phase 2 (1 week at max dose)

CONTACTS AND LOCATIONS:
Overall Officials: Eva G. Widerstrom-Noga, DDS PhD, Principal Investigator — VA Medical Center, Miami
Locations (1):
- VA Medical Center, Miami, Miami, Florida, United States

REFERENCES:
- [Result] Sindrup SH, Jensen TS. Efficacy of pharmacological treatments of neuropathic pain: an update and effect related to mechanism of drug action. Pain. 1999 Dec;83(3):389-400. doi: 10.1016/S0304-3959(99)00154-2. PMID 10568846
- [Result] Defrin R, Ohry A, Blumen N, Urca G. Characterization of chronic pain and somatosensory function in spinal cord injury subjects. Pain. 2001 Jan;89(2-3):253-63. doi: 10.1016/s0304-3959(00)00369-9. PMID 11166482
- [Result] Widerstrom-Noga EG, Felipe-Cuervo E, Yezierski RP. Chronic pain after spinal injury: interference with sleep and daily activities. Arch Phys Med Rehabil. 2001 Nov;82(11):1571-7. doi: 10.1053/apmr.2001.26068. PMID 11689978
- [Result] Tasmuth T, Hartel B, Kalso E. Venlafaxine in neuropathic pain following treatment of breast cancer. Eur J Pain. 2002;6(1):17-24. doi: 10.1053/eujp.2001.0266. PMID 11888224
- [Result] Westgren N, Levi R. Quality of life and traumatic spinal cord injury. Arch Phys Med Rehabil. 1998 Nov;79(11):1433-9. doi: 10.1016/s0003-9993(98)90240-4. PMID 9821906